CLINICAL TRIAL: NCT05004805
Title: COVID-19 Methylene Blue Antiviral Treatment
Acronym: COMBAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Irkutsk Scientific Center of the Siberian Branch of the Russian Academy of Sciences (Other Government)
Collaborators: Irkutsk State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COMBAT
Record Dates: First submitted 2021-08-11; First posted 2021-08-13 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Methylene Blue

STUDY DESIGN:
Intervention Model Description: Single-center, blind, randomized, controlled clinical trial.
Who Masked: Outcomes Assessor
Masking Description: Randomization by phone
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylene blue Arm (Experimental): The intervention is carried out in addition to the standard treatment. Administered Intervention is topical application of 0.02% Methylene blue solution in the form of repeated nasopharyngeal irrigation. The investigational drug is equipped with a spray nozzle to perform three administrations into both lower nasal passages. After three administrations on each side, it is recommended to take a deep breath so that the injected solution is distributed along the nasopharynx and oropharynx every 4 hours (5-6 times a day with a break for sleep). Duration is the period of stay of the subject, as long as there is no need for non-invasive or invasive mechanical ventilation. If the subject refuses further treatment in a hospital but does not withdraw consent to participate in the study, they should continue to take study drug after discharge from hospital, but not later than the date of the follow-up visit.
  Interventions: Drug: Methylene Blue
- Saline solution Arm (Placebo Comparator): The intervention is carried out in addition to the standard treatment. Adminestered Intervention is saline solution in the form of repeated nasopharyngeal irrigation. Dosage form, dosage, frequency and duration of intervention are the same.
  Interventions: Drug: Saline nasal spray

INTERVENTIONS:
Drug: Methylene Blue — MB administered topically as a 0.02% solution nasal spray in COVID-19 patients requiring hospitalization.
  Other Names: MB Spray
  Arms: Methylene blue Arm
Drug: Saline nasal spray — Saline administered topically as nasal spray in COVID-19 patients requiring hospitalization.
  Other Names: Placebo Spray
  Arms: Saline solution Arm

SUMMARY:
This is a pilot study of a single-center, blind, randomized, placebo-controlled, parallel-group study testing for the efficacy and safety of Methylene blue when administered topically as a 0.02% solution for nasopharyngeal and oropharyngeal irrigation in COVID-19 patients requiring hospitalization.

DETAILED DESCRIPTION:
Purpose of the study. To test the hypothesis that the topical application of 0.02% MB solution in the form of repeated nasopharyngeal irrigation will lead to an accelerated recovery compared to placebo, defined by the clinical, laboratory, and radiological improvement with a negative molecular test for SARS-CoV-2 by polymerase chain reaction (PCR). The main objective of the study is to demonstrate the effectiveness of 0.02% MB irrigation of the nasopharynx mucosa over placebo, alongside the standard treatment carried out in accordance with the Temporary Guidelines of "Prevention, Diagnosis, and Treatment of Novel Coronavirus Infection (COVID-19)", version 11 (May 7, 2021). Regarding the recovery of patients with COVID-19, this is defined as a negative PCR test result for the SARS-CoV-2 coronavirus in swabs from the nasopharynx and oropharynx on the 14th and 28th day after initiation of the experimental treatment.

A secondary objective of this study is to evaluate the additional efficacy and overall safety parameters, including saturation dynamics, C-reactive protein, D-dimer, CT signs of lung damage, dynamics of the National Early Warning Score (NEWS) 2 during treatment. Due to the pilot nature of this study, another goal is to calculate the effect based on the number of subjects per group for a future study.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 and over at the time of signing the informed consent.
2. The patient is willing and able to give written informed consent to participate in the study and follow the procedures specified in the protocol.
3. Diagnosed with COVID-19, confirmed by a PCR test positive for the SARS-CoV-2 coronavirus in smears from the nasopharynx and oropharynx.
4. Indications for hospitalization for COVID-19 treatment: a moderate condition that does not require oxygen support or low oxygen flow required through a nasal cannula or oxygen mask.
5. A urine test performed during screening, negative for pregnancy in women capable of childbearing.

Exclusion Criteria:

1. The need for non-invasive ventilation or high oxygen flow, or intubation of the trachea with artificial ventilation, or the use of vasopressors and/or extracorporeal membrane oxygenation at the time of assessment.
2. Decompensation of concomitant pathology, whose severity exceeds the severity of COVID-19 manifestations (for example, acute coronary syndrome, cerebral circulation disorders, acute surgical pathology requiring surgical intervention, bleeding independent of the localization, etc.).
3. Topical or systemic use of Methylene blue for any reasons at the time of evaluation or during the interval of 30 days before hospitalization.
4. Known intolerance or hypersensitivity to Methylene blue (indicated in the medical history of the patient).
5. Patients with a high probability of not surviving within the first 24 h of hospitalization, regardless of the treatment, as defined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
Recovery | Day 14 after randomization
  A negative PCR test result for the SARS-CoV-2 using nasopharyngeal and oropharyngeal swabs
Recovery | Day 28 after randomization
  A negative PCR test result for the SARS-CoV-2 using nasopharyngeal and oropharyngeal swabs

SECONDARY OUTCOMES:
Clinical responce | Day 28 after randomization
  Determined by the investigator
Overall therapeutic response | Day 28 after randomization
  The overall therapeutic response defined as a "general cure" or "treatment failure" and is calculated for each patient according to the patient's combination of clinical, radiological response, and PCR result.
Resolution rate | Day 28 after randomization
  The rate of resolution of fever, normalization of SpO2 (NEWS2), dynamics of target laboratory parameters (C-reactive protein, D-dimer)
Clinical responce FUV | Follow up visit, week 4 ± 3 days after discharge from the hospital
  Determined by the investigator
Overall therapeutic response FUV | Follow up visit, week 4 ± 3 days after discharge from the hospital
  The overall therapeutic response defined as a "general cure" or "treatment failure" and is calculated for each patient according to the patient's combination of clinical, radiological response, and PCR result.

CONTACTS AND LOCATIONS:
Locations (1):
- Irkutsk Regional Hospital, Irkutsk, Irkutsk Oblast, Russia